CLINICAL TRIAL: NCT04372381
Title: Supra-Annular vs. Annular ValvEs for Small Annuli (<= 23mm)
Brief Title: Supra-Annular vs. Annular ValvEs for Small Annuli
Acronym: SAVE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Marvin Eng (Other)
Collaborators: Corewell Health East (Other)
Responsible Party: Sponsor-Investigator, Marvin Eng, Associate Professor, Internal Medicine, University of Arizona
Organization: University of Arizona (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000164
Record Dates: First submitted 2020-04-27; First posted 2020-05-04 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Aortic Valve Stenosis; Implantation, Heart Valve Prosthesis
Keywords: Implantation, Heart Valve Prosthesis; aortic valve stenosis; transcatheter aortic valve replacement
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Intervention Model Description: Open-Label, Prospective randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Supra-Annular transcatheter heart valve (Active Comparator): Medtronic Evolut Pro Valve implantation
  Interventions: Device: Transcatheter aortic valve replacement (Edwards Sapien Ultra or Medtronic Evolut Pro
- Annular transcatheter heart valve (Active Comparator): Edwards Sapien 3 Ultra implantation
  Interventions: Device: Transcatheter aortic valve replacement (Edwards Sapien Ultra or Medtronic Evolut Pro

INTERVENTIONS:
Device: Transcatheter aortic valve replacement (Edwards Sapien Ultra or Medtronic Evolut Pro — Treatment of aortic valve stenosis using transcatheter aortic valve replacement

SUMMARY:
Open-label, prospective randomized comparison of Supra-annular valves (Medtronic Evolut Pro) vs. annular valves (Edwards Sapien Ultra) for small annuli (≤23 mm)

DETAILED DESCRIPTION:
Patient prothesis mis-match (PPM) remains a clinical dilemma in transcatheter aortic valve replacement (TAVR) and has been linked to higher rates of morbidity and mortality. Supra-annular self-expanding valves have been linked to lower gradients and lower rates of patient prosthesis mismatch versus annular valves but they have not been directly compared. Patients with small annuli are particularly vulnerable to PPM, therefore, the aprior hypothesis is that implantation of supra-annular valves for small annuli may show differences in PPM rates and outcomes when compared to annular valves.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic subjects with severe native aortic valve stenosis
* aortic valve annulus mean diameter ≤23 mm
* Patient meet commercial indication for transcatheter aortic valve replacement (TAVR)
* Institutional heart team determines that TAVR is appropriate
* Patient's anatomy is appropriate for either Medtronic Evolute or Edwards Sapien 3 Ultra

Exclusion Criteria:

* Subject unable or unwilling to provide informed consent
* Intended concurrent structural heart procedure (e.g. transcatheter mitral valve repair or replacement, left atrial appendage closure)
* Renal function precluding the administration of iodinated contrast (eGFR < 30ml/min/1.73m2). An exception to this exclusion criterion is made if the subject is established on renal replacement therapy and is therefore able to receive intravenous iodinated contrast media
* Pregnancy or intent on becoming pregnant prior to completion of all proctocol follow-up procedures
* Patients at high risk for coronary obstruction
* Patients with low-flow low gradient aortic valve stenosis
* patients at high risk for annular rupture with implantation of a balloon expandable valve

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-05-12 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint of patient prosthesis mismatch and >= moderate paravalvular regurgitation | 1 month

SECONDARY OUTCOMES:
VARC-2 30-day early safety and efficacy | 30 days
  All cause mortality stroke life-threatening bleeding acute kidney injury-stage 2 or 3 coronary artery obstruction major vascular complication valve-related dysfunction requiring repeat procedure NYHA class III or IV Requiring hospitalization for valve-related symptoms or worsening congestive heart failure
Pacemaker implantation | 30 days
  Clinical indication for permanent pacemaker insertion
Prosthetic Valve Dysfunction | 30 days and 1 year
  Mean aortic valve gradient >= 20 mmHg
  >= Moderate transvalvular aortic regurgitation Abnormal leaflet thickening Decreased leaflet mobility Leaflet thrombosis

CONTACTS AND LOCATIONS:
Overall Officials: Marvin Eng, MD, Principal Investigator — University of Arizona
Locations (3):
- United States (3):
  - Banner - University Medical Center, Phoenix campus, Phoenix, Arizona
  - Tucson Medical Center, Tucson, Arizona
  - Delray Medical Center, Delray Beach, Florida

IPD SHARING:
Plan to Share IPD: No